CLINICAL TRIAL: NCT06831955
Title: The LESLIE Trial: LifEStyle Intervention to Enhance Efficacy of Neoadjuvant Systemic Therapy in Patients With Triple Negative Breast Cancer
Brief Title: LifEStyle Intervention to Enhance Efficacy of Neoadjuvant Therapy in Patients With Triple Negative Breast Cancer
Acronym: LESLIE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); AZ Groeninge (Unknown); Jessa Ziekenhuis Hasselt (Unknown); UZ Gent, Belgium (Unknown); UZ Antwerpen (Unknown); Ziekenhuis ad Stroom, Antwerpen (Unknown); Institute Gustave Roussy Paris (Unknown); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S69524
Record Dates: First submitted 2024-12-05; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-10

CONDITIONS: Triple Negative Breast Cancer (TNBC), Early Setting
Keywords: Triple Negative Breast Cancer; Lifestyle Intervention; Neoadjuvant treatment; Fasting-Mimicking Diet; Exercise therapy; Pathological Complete Response
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: control arm (Active Comparator): SOC neoadjuvant therapy is based on the systemic treatment regimen described in the Keynote 522 trial, apart from some minor changes.
  Interventions: Drug: SOC
- Arm B: Intervention arm (Experimental): Next to the SOC, the lifestyle intervention (cyclic FMD and exercise) will be part of the treatment.
  Interventions: Other: Exercise Therapy; Dietary Supplement: Fasting-Mimicking Diet; Drug: SOC

INTERVENTIONS:
Other: Exercise Therapy — The exercise regimen consists of a non-linear aerobic exercise program of 3-4 sessions per week. During days of FMD no exercise will be prescribed.
  Arms: Arm B: Intervention arm
Dietary Supplement: Fasting-Mimicking Diet — The FMD is a plant-based, low-carbohydrate, low-caloric diet of 4 days , with the fourth day being the day of chemo/immunotherapy. A total of 6 FMD cycles will be administered over the treatment period of 20 weeks.
  Arms: Arm B: Intervention arm
Drug: SOC — Four cycles of an intravenous infusion of pembrolizumab (200 mg) once every 3 weeks plus paclitaxel (80 mg per square meter of body-surface area once weekly) plus carboplatin (at a dose based on an area under the concentration-time curve of 1.5 mg per milliliter per minute) once weekly in the first 12 weeks, followed by four cycles of epirubicin (90 mg per square meter) plus cyclophosphamide (600 mg per square meter) once every 2 weeks plus pembrolizumab 400mg every 6 weeks or pembrolizumab 200mg every 3 weeks in the subsequent 8 weeks.

SUMMARY:
LESLIE is a multicentric randomized controlled trial in patients with triple negative breast cancer receiving neoadjuvant chemo/immunotherapy (NAT). This trial investigates the hypothesis that adding a cyclic fasting-mimicking diet combined with exercise during the NAT improves the NAT's therapeutic efficacy, treatment tolerability and compliance, as well as improve quality of life.

DETAILED DESCRIPTION:
Leslie is a 2-arms randomized (2:1) Phase IIb clinical trial including 356 patients that will investigate whether combining a cyclic FMD-based intervention with exercise concomitant with neoadjuvant systemic therapy may have a beneficial effect on treatment response, survival, treatment tolerability and compliance, as well as quality of life of patients with TNBC. The neoadjuvant treatment will last for 21 weeks in both arms. Visits to the day clinic will be scheduled for administration of Standard of Care (SOC) in combination with 2-weekly visits to physiotherapists and online support of onco-dietician for patients from arm B.

The control group (arm A): SOC neoadjuvant therapy is based on the systemic treatment regimen described in the Keynote 522 trial, apart from some minor changes. It consists of four cycles of an intravenous infusion of pembrolizumab (200 mg) once every 3 weeks plus paclitaxel (80 mg per square meter of body-surface area once weekly) plus carboplatin (at a dose based on an area under the concentration-time curve of 1.5 mg per milliliter per minute) once weekly in the first 12 weeks, followed by four cycles of epirubicin (90 mg per square meter) plus cyclophosphamide (600 mg per square meter) once every 2 weeks plus pembrolizumab 400mg every 6 weeks or pembrolizumab 200mg every 3 weeks in the subsequent 8 weeks. All treatments after surgery will be administered according to the institutional guidelines.

The interventional group (arm B): Next to the SOC, the lifestyle intervention (cyclic FMD and exercise) will be part of the treatment. The FMD is a plant-based, low-carbohydrate, low-caloric diet of 4 days , with the fourth day being the day of chemo/immunotherapy. A total of 6 FMD cycles will be administered over the treatment period of 20 weeks. The exercise regimen consists of a non-linear aerobic exercise program of 3-4 sessions per week. During days of FMD no exercise will be prescribed.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a biopsy-confirmed diagnosis of stage II-III TNBC

  1. Patients with tumor stage T1cN1-2, T2N0-N2, T3N0-N2, T4N0-N2
  2. ER and PR negative is defined as an absent or minimal (≤10%) expression of oestrogen and progesterone receptors and absence of HER2 protein over-expression per ASCO/CAP-guidelines
  3. All histological subtypes are eligible, including but not limited to invasive breast cancer of no special type (NST) , invasive lobular carcinoma (ILC) etc
* WHO/ECOG performance status of grade 0-1
* The participant is able to perform a CPET test (cardiopulmonary exercise testing)
* Body mass index ≥ 18.5 kg/m²
* Pregnant or breastfeeding women
* Presence of adequate bone marrow and organ function
* HbA1c <10%

Exclusion Criteria:

* had a treatment with any of the following:

  1. any other chemotherapy, immunotherapy or anticancer agents within 5 years of the first dose of study treatment
  2. injectable hypoglycemics 2. have not have recovered adequately from the toxicity and/or complications from a surgical intervention prior to starting therapy
* prior systemic treatment for breast cancer or other malignancies within 5 years of treatment enrollment, except for adequately treated basal cell or squamous skin cancer or in situ cervical cancer. Other malignancies diagnosed more than 5 years before the diagnosis of breast cancer must have been radically treated without evidence of relapse at the moment of patient enrollment in the trial.
* has a history of an additional malignancy that is progressing or that has required active treatment in the 5 years prior to breast cancer diagnosis. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Prior treatment with anthracyclines
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
* Has any disorder, which in the Investigator's opinion might jeopardize the participant's safety or compliance with the protocol
* Has, as judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV). Screening for chronic conditions is not required
* Active autoimmune diseases requiring systemic treatments
* Patients with type 1 diabetes mellitus
* History of alcohol use disorder (DSM-5)
* History of eating disorder (DSM-5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Surgical specimen (at the time of surgery)
  pCR, ypT0/Tis ypN0: no invasive residual disease in breast or regional lymph nodes; residual in situ disease allowed

SECONDARY OUTCOMES:
Adherence and compliance to FMD | 20 weeks, in case of dose delays up to 30 weeks
  Adherence is defined as the ratio of how many days the patient complies to the FMD (without 2 minor or 1 major deviation), divided by the in total 24 planned days of FMD. Compliance will be measured at the end of each FMD cycle based on the incidence of minor and major deviations from the prescribed dietary regimen.
Adherence and compliance to exercise therapy | 20 weeks, in case of dose delays up to 30 weeks
  Exercise attendance is calculated as the number of training sessions attended divided by the total 75 planned sessions. Compliance is calculated based on the relative dose intensity (RDI). Relative dose intensity (RDI) is defined as the ratio of total completed to total planned cumulative dose, expressed as a percentage.
Adverse Event profile | Following completion of the NAT, subjects will be followed for 30 days for AEs, SAEs will be collected for 90 days after completion of NAT. An exception is made for heart failure which will be collected till 1 year after NAT.
  The type, incidence, severity (as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0), seriousness, time till onset and duration of Adverse Events (AEs)/SAEs, immune-related AEs and any laboratory abnormalities
Systemic Treatment Completion | 20 weeks, in case of dose delays up to 30 weeks
  RDI is defined as the amount of drug administered per unit of time (=delivered total dose in mg/m2 divided by actual time used to complete treatment in a number of weeks) as a fraction of the standard amount of drug per unit of time (=standard total dose in mg/m2 divided by standard time to complete treatment in a number of weeks)
Event-Free Survival (EFS) at 3 years | From the date of randomization to the first documentation of progressive disease or patient death, assessed up to 36 months
  at 3 years is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause. Patients without documented event at the time of the analysis will be censored at the date of the last follow-up
Distant Metastasis-Free Survival at 3 years | From surgery to the occurrence of distant metastases or patient death, assessed up to 36 months
  is defined as the time from randomization to the occurrence of distant metastasis or death. Patients without documented event at the time of the analysis will be censored at the date of the last follow-up.
Residual Cancer Burden | Surgical specimen (at the time of surgery)
  Residual Cancer Burden (RCB) continuous score and categories calculated using the classification by Symmans et al with RCB-0 (pCR [ypT0/Tis ypN0]), RCB-I (minimal residual disease), RCB-II (moderate residual disease), and RCB-III (extensive residual disease or progression on neoadjuvant therapy). In the breast the primary tumor beds' dimensions and overall cancer cellularity is considered, including the percentage of cancer that is in situ disease in tumor bed. For lymph nodes the number of positive lymph nodes and the size of the largest metastatic deposit is used.
Quality of life (QoL) | From the date of randomization up to 36 months
  Quality of life (QoL): as assessed using the European Organisation for Research and Treatment of Cancer (EORTC) questionnaires EORTC-QLQ-C30 and EORTCQLQ- BR42. The questionnaires will be filled in at baseline, at C8 and C14, week before surgery and at 3 months, 6 months, 1 year, 2 years and 3 years postoperative.
Body Composition | From the date of randomization up to 36 months
  as evaluated with weekly bioimpedance measurements (fat-free mass, fat mass, phase angle, extracellular mass-to-body cell mass ratio (ECM/BCM), total body water and intracellular water). This scale is designed following the ISO 13 485 and the Medical Device Regulation (MDR) guidelines. After com
Fatigue | From the date of randomization up to 36 months
  Fatigue: as assessed using the FACIT-Fatigue v4.0 questionnaire. The questionnaire will be filled in at baseline, at C8 and C14, week before surgery and at 3 months, 6 months, 1 year, 2 years and 3 years postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Desmedt, PhD, Principal Investigator — KU Leuven; Ann Smeets, MD, PhD, Principal Investigator — UZ Leuven
Locations (10):
- Belgium (10):
  - UZ Antwerpen, Antwerp
  - Ziekenhuis aan de Stroom, Antwerp
  - Cliniques universitaires Saint-Luc (UCLouvain), Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
  - Jessa Ziekenhuis Hasselt, Hasselt
  - AZ Groeninge, Kortrijk
  - University Hospital Leuven, Leuven
  - Centre Hospitalier Universitaire (CHU) UCL Liège, Liège
  - Centre Hospitalier Universitaire (CHU) UCL Namur, Namur

IPD SHARING:
Plan to Share IPD: No